CLINICAL TRIAL: NCT03088813
Title: RESILIENT: A Randomized, Open Label Phase 3 Study of Irinotecan Liposome Injection (ONIVYDE®) Versus Topotecan in Patients With Small Cell Lung Cancer Who Have Progressed on or After Platinum-based First-Line Therapy
Brief Title: Study of Irinotecan Liposome Injection (ONIVYDE®) in Patients With Small Cell Lung Cancer
Acronym: RESILIENT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ipsen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MM-398-01-03-04; 2017-004261-26 (EudraCT Number)
Record Dates: First submitted 2017-03-09; First posted 2017-03-23 (Actual); Results first posted 2023-10-17 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2025-02

CONDITIONS: Small Cell Lung Cancer
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — irinotecan sucrosofate; Topotecan

STUDY DESIGN:
Masking Description: Open Label
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Part 1: Experimental Arm, dose level 1 (Experimental): Irinotecan liposome injection
  Interventions: Drug: Irinotecan liposome injection
- Part 1: Experimental Arm, dose level 2 (Experimental): Irinotecan liposome injection
  Interventions: Drug: Irinotecan liposome injection
- Part 2: Experimental Arm (Experimental): Irinotecan liposome injection
  Interventions: Drug: Irinotecan liposome injection
- Part 2: Control Arm (Active Comparator): Topotecan
  Interventions: Drug: Topotecan

INTERVENTIONS:
Drug: Irinotecan liposome injection — IV
  Other Names: ONIVYDE®
  Arms: Part 1: Experimental Arm, dose level 1; Part 1: Experimental Arm, dose level 2; Part 2: Experimental Arm
Drug: Topotecan — IV
  Arms: Part 2: Control Arm

SUMMARY:
A randomized, open label phase 3 study of irinotecan liposome injection (ONIVYDE®) versus topotecan in patients with small cell lung cancer who have progressed on or after platinum-based first-line therapy

The study was conducted in two parts:

1. Dose determination of irinotecan liposome injection
2. A randomized, efficacy study of irinotecan liposome injection versus topotecan

DETAILED DESCRIPTION:
The study was conducted in two parts:

Part 1: Open-label dose-finding study of irinotecan liposome injection. 30 patients were planned to be enrolled.

Part 1 Primary Objectives:

* Describe the safety and tolerability of irinotecan liposome injection monotherapy administered every 2 weeks
* Determine the optimal irinotecan liposome injection monotherapy dose for Part 2 of this study

Part 2: A randomized, efficacy study of irinotecan liposome injection versus intravenous (IV) topotecan.

Approximately 450 patients were planned to be enrolled in part 2.

Part 2 objectives: To compare overall survival following treatment with irinotecan liposome injection with overall survival following treatment with IV topotecan.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age.
* Able to understand and provide an informed consent
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
* Life expectancy >12 weeks
* Histopathologically or cytologically confirmed small cell lung cancer
* Evaluable disease as defined by RECIST Version 1.1 guidelines (patients with non measurable lesions only are eligible).
* Radiologically confirmed progression on or after first-line platinum based chemotherapy (carboplatin or cisplatin), or chemo-radiation including platinum-based chemotherapy for treatment of limited or extensive stage Small Cell Lung Cancer (SCLC). In addition to platinum-based regimen, one line of immunotherapy as monotherapy or in combination, in first or in second line setting is allowed.
* Recovered from the effects of any prior chemotherapy, surgery, radiotherapy or other anti-neoplastic therapy (recovered to Grade 1 or better, with the exception of alopecia, peripheral neuropathy, or ototoxicity).
* Adequate bone marrow reserves
* Adequate hepatic function
* Adequate renal function
* Electrocardiogram during the Screening period without any clinically significant findings, per investigator's assessment
* Patients with certain types of asymptomatic CNS metastases that meet ALL the following criteria are eligible.

  1. Patients with asymptomatic CNS metastases prior to enrollment
  2. Prior radiation for CNS metastatic disease is completed ≥4 weeks prior to enrollment
  3. CNS metastases that are stable or have decreased according to the post radiation follow-up scan that is conducted at least 4 weeks after completion of radiation treatment for CNS lesion.
  4. Patients have discontinued corticosteroids or are on stable low-dose steroids (prednisone or equivalent 10 mg daily or less) for at least 1 week after completion of radiation for CNS lesion prior to enrollment.

Exclusion Criteria

* Any medical or social condition deemed by the Investigator to be likely to interfere with a patient's ability to sign informed consent, cooperate and participate in the study, or interfere with the interpretation of the results
* Pregnant or breast feeding;
* Patients with large cell neuroendocrine lung carcinoma.
* Patients who have received prior topoisomerase I inhibitor treatment, retreatment with platinum-based regimen, antibody-drug conjugates or molecular targeted agents, more than one line of immunotherapy, or any other additional regimen of prior cytotoxic chemotherapy.
* Patients with the symptomatic Central Nervous System (CNS) metastasis and/or who have developed new or progressive brain metastasis within 3 months following prophylactic and/or therapeutic cranial radiation (whole brain stereotactic radiation).
* Patients with carcinomatous meningitis.
* Unable to discontinue the use of strong CYP3A4 or UGT1A1 inhibitors at least 1 week or strong CYP3A4 inducers at least 2 weeks prior to receiving the first dose of irinotecan liposome injection.
* Have a previous or concurrent cancer that is distinct in primary (non-pulmonary) site or SCLC histology
* Investigational therapy administered within 4 weeks, or within a time interval less than at least 5 half-lives of the investigational agent, whichever is less, prior to the first scheduled day of dosing in this study.
* Severe cardiovascular and pulmonary diseases
* New York Heart Association Class III or IV congestive heart failure, ventricular arrhythmias, or uncontrolled blood pressure.
* Active infection
* Known hypersensitivity to any of the components of irinotecan liposome injection, other liposomal products, or topotecan.
* Clinically significant gastrointestinal disorder including hepatic disorders, bleeding, inflammation, occlusion, or diarrhea > grade 1.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 491 (Actual)
Dates: Start 2018-04-25 (Actual); Primary Completion 2022-02-08 (Actual); Study Completion 2023-07-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ipsen Medical Director, Study Director — Ipsen
Locations (118):
- United States (22):
  - National Jewish Health, Denver, Colorado
  - Rocky Mountain Cancer Centers, Denver, Colorado
  - Florida Cancer Specialists (South Region), Fort Myers, Florida
  - Florida Cancer Specialists, St. Petersburg, Florida
  - Northwest Georgia Oncology Centers, Marietta, Georgia
  - Cancer Treatment Centers of America-Georgia, Newnan, Georgia
  - Illinois Cancer Care, PC, Peoria, Illinois
  - Southern Maine Health Care, Biddeford, Maine
  - University of Maryland Medical Group, Baltimore, Maryland
  - Henry Ford Hospital, Detroit, Michigan
  - Cancer & Hematology Centers of Western Michigan, Grand Rapids, Michigan
  - Sparrow Regional Cancer Center, Lansing, Michigan
  - Roswell Park Cancer Institute, Buffalo, New York
  - North Shore Hematology Oncology Associates, PC, East Setauket, New York
  - Case Western Reserve University, Cleveland, Ohio
  - Tri County Hematology & Oncology Associates, Inc, Massillon, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Charleston Hematology Oncology Associates, PA, Charleston, South Carolina
  - Greenville Hospital System University Medical Center, Greenville, South Carolina
  - Tennessee Oncology, Nashville, Tennessee
  - MultiCare Health System Institute for Research and Innovation, Spokane, Washington
  - Summit Cancer Treatment Center, Spokane, Washington
- Australia (4):
  - Border Medical Oncology Research Unit, Albury, New South Wales
  - South West Healthcare, Warrnambool, Victoria
  - Southern Medical Day Care Centre, Wollongong
  - Princess Alexandra Hospital, Woolloongabba
- Belgium (4):
  - AZ Klina, Brasschaat
  - UZ Leuven, Leuven
  - Centre Hospitalier de l'Ardenne, Libramont
  - AZ Sint-Maarten, Mechelen
- Brazil (8):
  - Hospital de Cancer de Barretos, Fundacoa Pio X II, Barretos
  - Hospital de Caridade de Ijuí, Ijuí
  - Oncobio Servicos de Saude, Nova Lima
  - HGB - Hospital Giovanni Battista - Mãe de Deus Center, Porto Alegre
  - Hospital Nossa Senhora da Conceição, Porto Alegre
  - INCA - Instituto Nacional de Câncer, Rio de Janeiro
  - CEPHO - Centro de Estudos e Pesquisas de Hematologia e Oncologia, Santo André
  - Fundação Faculdade Regional de Medicina de São José do Rio Preto, São José do Rio Preto
- China (9):
  - Beijing Cancer Hospital, Beijing
  - The First Affiliated Hospital of Bengbu Medical College, Bengbu
  - The First Hospital of Jilin University, Changchun
  - West China Hospital, Sichuan University, Chengdu
  - Guangdong Provincial People's Hospital, Guangzhou
  - Zhejiang Cancer Hospital, Hangzhou
  - Tongji Hospital, Hubei
  - Linyi Cancer Hospital, Linyi
  - Henan Cancer Hospital, Zhengzhou
- France (4):
  - CHU Brest - Hôpital Morvan, Brest
  - Hôpital Nord - CHU Marseille, Marseille
  - Institut de Cancérologie de la Loire, Saint-Priest-en-Jarez
  - Centre Hospitalier de Saint-Quentin, Saint-Quentin
- Germany (4):
  - Universitaetsklinikum Freiburg, Freiburg im Breisgau
  - Evangelisches Krankenhaus Hamm GmbH, Hamm
  - Universitaetsklinikum Heidelberg, Heidelberg
  - Pius-Hospital Oldenburg, Oldenburg
- Hungary (5):
  - Semmelweis Egyetem, Budapest
  - Bekes Megyei Kozponti Korhaz Pandy Kalman Tagkorhaza, Gyula
  - Jasz-Nagykun-Szolnok Megyei Hetenyi Geza Korhaz-Rendelointezet, Szolnok
  - Tudogyogyintezet Torokbalint, Törökbálint
  - Zala Megyei Szent Rafael Korhaz, Zalaegerszeg
- Italy (3):
  - Istituto Scientifico Romagnolo Per Lo Studio e La Cura Dei Tumori, Meldola
  - Fondazione IRCCS Istituto Nazionale dei Tumori, Milan
  - Azienda Sanitaria Universitaria Integrata di Udine, Udine
- Poland (5):
  - KO-MED Centra Kliniczne Biala Podlaska, Biała Podlaska
  - Szpitale Pomorskie spółka z ograniczoną odpowiedzialnością, Gdynia
  - SP Zespol Gruzlicy i Chorob Pluc w Olsztynie, Olsztyn
  - Przychodnia Med-Polonia Sp. z o.o., Poznan
  - Szpital Kliniczny Przemienienia Panskiego Uniwersytetu Medycznego im. Karola Marcinkowskiego, Poznan
- Romania (6):
  - S.C Gral Medical S.R.L, Bucharest
  - Institutul Oncologic "Prof. Dr. Ion Chiricuta" Cluj-Napoca, Cluj-Napoca
  - S.C Medisprof S.R.L, Cluj-Napoca
  - S.C Centrul de Oncologie Sf. Nectarie S.R.L, Craiova
  - S.C Radiotherapy Center Cluj S.R.L, Floreşti
  - Oncomed SRL, Timișoara
- Russia (6):
  - SBIH of Arkhangelsk region "Arkhangelsk Clinical Oncological Dispensary", Arkhangelsk
  - "VitaMed" LLC, Moscow
  - BHI of Omsk region "Clinical Oncology Dispensary", Omsk
  - SBHI of Kaluga Region "Kaluga regional clinical oncology dispensary", Saint Petersburg
  - SPb SBIH "City Clinical Oncological Dispensary", Saint Petersburg
  - SBIH of Yaroslavl region "Regional Clinical Oncological Hospital", Yaroslavl
- Serbia (5):
  - Clinical Center "Bezanijska kosa", Belgrade
  - Clinical Center Kragujevac, Belgrade
  - Oncomed System, Belgrade
  - Institute for Pulmonary Diseases of Vojvodina, Kamenitz
  - General Hospital Uzice, Užice
- South Korea (4):
  - Chungbuk National University Hospital, Cheongju-si
  - Asan Medical Center, Seoul
  - The Catholic University of Korea, Seoul St. Mary's Hospital, Seoul
  - The Catholic University of Korea, St. Vincent's Hospital, Suwon
- Spain (8):
  - ICO l'Hospitalet - Hospital Duran i Reynals, L'Hospitalet de Llobregat, Barcelona
  - Hospital General Universitario de Alicante, Alicante
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital General Universitario Gregorio Marañon, Madrid
  - Hospital Regional Universitario de Malaga, Málaga
  - Hospital Universitario Virgen del Rocio, Seville
  - Hospital Universitari i Politecnic La Fe, Valencia
- Taiwan (5):
  - Changhua Christian Hospital, Changhua
  - Kaohsiung Chang Gung Memorial Hospital, Kaohsiung City
  - National Taiwan University Hospital, Taipei
  - Tri-Service General Hospital, Taipei
  - Chang Gung Memorial Hospital, Linkou, Taoyuan District
- Turkey (Türkiye) (6):
  - Baskent University Adana Application and Research Center, Adana
  - Trakya University Medical Faculty, Edirne
  - Istanbul Medeniyet Uni Goztepe Training&Res Hosp, Istanbul
  - Istanbul University Cerrahpasa - Cerrahpasa Medical Faculty, Istanbul
  - Inonu Uni. Med. Fac., Malatya
  - Namik Kemal University, Tekirdağ
- Ukraine (10):
  - CI Chernivtsi RC Oncological Dispensary, Chernivtsi
  - CI Dnipropetrovsk CMCH #4 of Dnipropetrovsk RC Dept of Chemotherapy SI Dnipropetrovsk MA of MOHU, Dnipro
  - Communal Non-profit Enterprise Regional Center of Oncology, Kharkiv
  - Communal Enterprise Kremenchuk Regional Oncology Dispensary of Poltava Regional Council, Kremenchuk
  - CI Kryvyi Rih Oncological Dispensary of DRC, Kryvyi Rih
  - Treatment-Prevention Institution Volyn Regional Oncological Dispensary, Lutsk
  - Odesa Regional Oncologic Dispensary, Odesa
  - RCI Sumy Regional Clinical Oncological Dispensary, Sumy
  - CCCH City Oncological Center SHEI Uzhgorod NU, Uzhhorod
  - Medical Clinic Innovacia, LLC, Vyshhorod

REFERENCES:
- [Derived] Spigel DR, Dowlati A, Chen Y, Navarro A, Yang JC, Stojanovic G, Jove M, Rich P, Andric ZG, Wu YL, Rudin CM, Chen H, Zhang L, Yeung S, Benzaghou F, Paz-Ares L, Bunn PA; RESILIENT Trial Investigators. RESILIENT Part 2: A Randomized, Open-Label Phase III Study of Liposomal Irinotecan Versus Topotecan in Adults With Relapsed Small Cell Lung Cancer. J Clin Oncol. 2024 Jul 1;42(19):2317-2326. doi: 10.1200/JCO.23.02110. Epub 2024 Apr 22. PMID 38648575
- [Derived] Paz-Ares L, Spigel DR, Chen Y, Jove M, Juan-Vidal O, Rich P, Hayes T, Calderon VG, Caro RB, Navarro A, Dowlati A, Zhang B, Moore Y, Yao X, Kokhreidze J, Ponce S, Bunn PA. RESILIENT part 1: a phase 2 dose-exploration and dose-expansion study of second-line liposomal irinotecan in adults with small cell lung cancer. Cancer. 2022 May 1;128(9):1801-1811. doi: 10.1002/cncr.34123. Epub 2022 Feb 23. PMID 35195913
- See also: Lay language results summary — https://www.ipsen.com/websites/ipsen_com_v2/wp-content/uploads/2024/11/08172330/MM-398-01-03-04-lay-results-summary.pdf

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This Phase III, 2-part (Part 1: [open-label, single-arm dose evaluation period] and Part 2 [randomized, open-label period]) study was conducted in participants with small cell lung cancer (SCLC) who progressed on or after platinum-based first-line therapy at 11 sites for Part 1 and 116 sites for Part 2 in the USA, Europe, Asia, Australia, Turkey and Brazil. First participant was enrolled on 25 April 2018 and primary analysis data cut-off (DCO) date was 08 February 2022 for Part 2.
Pre-assignment Details: Each part consisted of screening stage (up to 28 days), treatment/active follow-up stage, and a long-term monthly follow-up stage. A total of 30 participants in Part 1 received study treatment and 461 participants in Part 2 were randomized to receive study treatment in this study.
Groups:
- Part 1: Irinotecan Liposome Injection 85 Milligrams/Meter Square (mg/m^2): Participants received irinotecan liposome injection 85 mg/m^2 intravenously (i.v.) over 90 minutes every 2 weeks in a 6-week cycle until disease progression (PD), death, unacceptable study treatment-related toxicity or withdrawal of consent.
- Part 1: Irinotecan Liposome Injection 70 mg/m^2: Participants received irinotecan liposome injection 70 mg/m^2 i.v. over 90 minutes every 2 weeks in a 6-week cycle until PD, death, unacceptable study treatment-related toxicity or withdrawal of consent.
- Part 2: Irinotecan Liposome Injection 70 mg/m^2: Eligible participants received irinotecan liposome injection 70 mg/m^2 i.v. over 90 minutes, every 2 weeks in a 6-week cycle until PD, death, unacceptable study treatment-related toxicity or withdrawal of consent.
- Part 2: Topotecan 1.5 mg/m^2: Eligible participants received topotecan 1.5 mg/m^2 i.v. over 30 minutes daily for 5 consecutive days, every 3 weeks in a 6-week cycle until PD, death, unacceptable study treatment-related toxicity or withdrawal of consent.
Period: Part 1: Dose Evaluation (Up to Week 172)
Arm/Group | Part 1: Irinotecan Liposome Injection 85 Milligrams/Meter Square (mg/m^2) | Part 1: Irinotecan Liposome Injection 70 mg/m^2 | Part 2: Irinotecan Liposome Injection 70 mg/m^2 | Part 2: Topotecan 1.5 mg/m^2
Started | 5 | 25 | 0 | 0
Completed | 5 | 24 | 0 | 0
Not Completed | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 0
Period: Part 2: Randomized Study (Upto Week 197)
Arm/Group | Part 1: Irinotecan Liposome Injection 85 Milligrams/Meter Square (mg/m^2) | Part 1: Irinotecan Liposome Injection 70 mg/m^2 | Part 2: Irinotecan Liposome Injection 70 mg/m^2 | Part 2: Topotecan 1.5 mg/m^2
Started | 0 | 0 | 229 | 232
Completed | 0 | 0 | 202 | 211
Not Completed | 0 | 0 | 27 | 21
Not completed — Protocol Violation | 0 | 0 | 1 | 0
Not completed — Investigator decision | 0 | 0 | 2 | 2
Not completed — Lost to Follow-up | 0 | 0 | 3 | 4
Not completed — Withdrawal by Subject | 0 | 0 | 18 | 14
Not completed — Screen failure | 0 | 0 | 0 | 1
Not completed — Other | 0 | 0 | 3 | 0

BASELINE CHARACTERISTICS:
Population: Part 1: Safety population included all enrolled participants who were treated with at least 1 dose of irinotecan liposome injection. Part 2: Intent-to-Treat (ITT) population included all randomized participants.
Groups:
- Part 1: Irinotecan Liposome Injection 85 mg/m^2: Participants received irinotecan liposome injection 85 mg/m^2 i.v. over 90 minutes every 2 weeks in a 6-week cycle until PD, death, unacceptable study treatment-related toxicity or withdrawal of consent.
- Total: Total of all reporting groups
Arm/Group | Part 1: Irinotecan Liposome Injection 85 mg/m^2 | Part 1: Irinotecan Liposome Injection 70 mg/m^2 | Part 2: Irinotecan Liposome Injection 70 mg/m^2 | Part 2: Topotecan 1.5 mg/m^2 | Total
Number analyzed (Participants) | 5 | 25 | 229 | 232 | 491
Age, Customized [Count of Participants; unit: Participants]
  <65 years | 4 | 18 | 128 | 151 | 301
  >=65 years | 1 | 7 | 101 | 81 | 190
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 16 | 79 | 69 | 166
  Male | 3 | 9 | 150 | 163 | 325
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 1 | 1
  Asian | 0 | 0 | 37 | 36 | 73
  Black or African American | 0 | 0 | 4 | 4 | 8
  White | 5 | 25 | 184 | 182 | 396
  Not Reported | 0 | 0 | 4 | 9 | 13
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 2 | 6 | 9 | 17
  Not Hispanic or Latino | 5 | 20 | 214 | 218 | 457
  Not Reported/Unknown | 0 | 3 | 9 | 5 | 17

OUTCOME MEASURES:

1. Primary Outcome: Part 1: Number of Participants With Treatment-Emergent Adverse Events (TEAEs) and Treatment-Emergent Serious Adverse Events (SAEs)
Description: An adverse event (AE) was any untoward medical occurrence in a participant following or during exposure to a study treatment, whether or not causally related to the study treatment. An undesirable medical condition could be symptoms, signs or abnormal results of an investigation. An SAE was any AE that: resulted in death; was life-threatening; required hospitalization or prolongation of existing hospitalization; resulted in persistent or significant disability or incapacity; resulted in congenital anomaly or birth defect; or was medically important. A TEAE was any AE that occurred or worsened on or after the day of first dose of study treatment and within 30 days after discontinuation of study treatment.
Time Frame: The TEAEs were reported from the time of first study treatment administration (Day 1) up to 30 days after the date of last study treatment administration, approximately 680 days
Population: Part 1: Safety population included all enrolled participants who were treated with at least 1 dose of irinotecan liposome injection.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: Irinotecan Liposome Injection 85 mg/m^2 | Part 1: Irinotecan Liposome Injection 70 mg/m^2
Number analyzed (Participants) | 5 | 25
Participants
  Any TEAE | 5 | 25
  Serious TEAEs | 4 | 9

2. Primary Outcome: Part 1: Number of Participants With Dose-Limiting Toxicities (DLT)
Description: A TEAE was considered as DLT if it occurred during the safety evaluation period (i.e. first 28 days of treatment or 14 days after the second dose of study treatment if there was a treatment delay due to non-DLT related reasons) and were deemed related to the study treatment by the investigator. The determination of whether an Adverse Event was considered a Dose Limiting Toxicity was made by the Safety Review Committee (SRC) comprising the Part 1 Investigators and the Medical Monitor(s) of the Sponsor.
Time Frame: From the start of the first study treatment administration (Day 1) up to 14 days after the second dose of study treatment administration, a maximum of 42 days
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: Irinotecan Liposome Injection 85 mg/m^2 | Part 1: Irinotecan Liposome Injection 70 mg/m^2
Number analyzed (Participants) | 5 | 25
Participants | 4 | 2

3. Primary Outcome: Part 2: Overall Survival (OS)
Description: The OS was defined as the time from randomization date to the date of death from any cause. In the absence of confirmation of death, survival time was censored at the last date the participant was known to be alive. The OS was calculated using Kaplan-Meier technique. Following end of treatment participant and/or family was contacted by telephone every month to assess vital status.
Time Frame: From date of randomization (within 7 days before start of study treatment) until death. Assessed up to Part 2 primary analysis DCO date of 08 February 2022 (approximately 900 days)
Population: Part 2: The ITT population included all randomized participants.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Part 2: Irinotecan Liposome Injection 70 mg/m^2 | Part 2: Topotecan 1.5 mg/m^2
Number analyzed (Participants) | 229 | 232
months | 7.92 [6.87 to 9.23] | 8.31 [7.33 to 9.13]
Statistical Analysis 1: Comparison: Part 2: Irinotecan Liposome Injection 70 mg/m^2 vs Part 2: Topotecan 1.5 mg/m^2; Test type: Other; p = 0.3094, Stratified log-rank test; From stratified log-rank test, stratified by corrected region and corrected platinum sensitivity; Hazard Ratio (HR) = 1.11, 95% CI 2-sided [0.90 to 1.37] — The associated HR and two-sided 95% Confidence Interval (CI) were estimated using stratified Cox proportional hazards model, stratified by corrected region and corrected platinum sensitivity

4. Secondary Outcome: Part 1: Objective Response Rate (ORR)
Description: The ORR was defined as the percentage of participants with a best overall response (BOR) characterized as either a complete response (CR) or partial response (PR) recorded from date of first dose of study treatment until documented PD or death. ORR analysis was based on BOR using RECIST v1.1 per investigator assessment. Per RECIST v1.1, CR is disappearance of all target lesions; PR is >=30% decrease in the sum of the longest diameter of target lesions; and overall response = CR + PR. Per protocol, participants had computed tomography (CT)-scans and brain magnetic resonance imaging (MRI) every 6 weeks to measure tumor lesion size. This was continued throughout treatment until PD or commencement of new anti-neoplastic therapy.
Time Frame: RECIST assessments performed at Baseline (within 28 days before start of study treatment), every 6 weeks post first dose and treatment pause, 30 days after discontinuation of study treatment, then every month thereafter, approximately maximum of 1177 days
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Part 1: Irinotecan Liposome Injection 85 mg/m^2 | Part 1: Irinotecan Liposome Injection 70 mg/m^2
Number analyzed (Participants) | 5 | 25
percentage of participants | 40 [5.27 to 85.34] | 44 [24.40 to 65.07]

5. Secondary Outcome: Part 1: Progression-Free Survival (PFS)
Description: The PFS was defined as time from first dose of study treatment to the first documented objective PD using RECIST v1.1 or death due to any cause, whichever occurs first. Per RECIST 1.1, progression is defined as at least 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions. The PFS was calculated using Kaplan-Meier technique. Per protocol, participants had CT-scans and brain MRI every 6 weeks to measure tumor lesion size. This was continued throughout treatment until PD or commencement of new anti-neoplastic therapy.
Time Frame: as for outcome 4
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Part 1: Irinotecan Liposome Injection 85 mg/m^2 | Part 1: Irinotecan Liposome Injection 70 mg/m^2
Number analyzed (Participants) | 5 | 25
months | 4.19 [1.58 to NA] — Upper limit of CI was not estimable due to insufficient number of participants with events at study closure. | 3.98 [2.69 to 4.24]

6. Secondary Outcome: Part 1: OS
Description: The OS was defined as the time from first dose of study treatment to the date of death from any cause. In the absence of confirmation of death, survival time was censored at the last date the participant was known to be alive. The OS was calculated using Kaplan-Meier technique. Following end of treatment participant and/or family was contacted by telephone every month to assess vital status.
Time Frame: From Baseline (Day 1) until death. Assessed up to Part 1 DCO date of 11 August 2021 (approximately 1177 days)
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Part 1: Irinotecan Liposome Injection 85 mg/m^2 | Part 1: Irinotecan Liposome Injection 70 mg/m^2
Number analyzed (Participants) | 5 | 25
months | 10.84 [0.99 to NA] — Upper limit of CI was not estimable due to insufficient number of participants with events at study closure. | 8.08 [5.16 to 9.82]

7. Secondary Outcome: Part 2: PFS
Description: The PFS was defined as time from randomization to first documented objective PD using RECIST 1.1 (or response assessment in neuro-oncology brain metastases [RANO-BM] criteria for central nervous system [CNS] lesions) as assessed by blinded independent central review (BICR) or death due to any cause, whichever occurred first. Per RECIST 1.1, progression is defined as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions. The PFS was calculated using Kaplan-Meier technique. Per protocol, participants had CT-scans and brain MRI every 6 weeks to measure tumor lesion size. This was continued throughout treatment until PD or commencement of new anti-neoplastic therapy.
Time Frame: RECIST assessments performed at Baseline (within 28 days before start of study treatment), every 6 weeks post first dose and treatment pause, 30 days after discontinuation of study treatment, then every month thereafter, approximately maximum of 900 days
Population: Part 2: The ITT population included all randomized participants.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Part 2: Irinotecan Liposome Injection 70 mg/m^2 | Part 2: Topotecan 1.5 mg/m^2
Number analyzed (Participants) | 229 | 232
months | 4.01 [2.96 to 4.17] | 3.25 [2.79 to 4.14]
Statistical Analysis 1: Comparison: Part 2: Irinotecan Liposome Injection 70 mg/m^2 vs Part 2: Topotecan 1.5 mg/m^2; Test type: Other; p = 0.7053, Stratified log-rank test — From stratified log-rank test, stratified by corrected region and corrected platinum sensitivity; Hazard Ratio (HR) = 0.96, 95% CI 2-sided [0.77 to 1.20] — The associated HR and two-sided 95% CI were estimated using stratified Cox proportional hazards model, stratified by corrected region and corrected platinum sensitivity

8. Secondary Outcome: Part 2: ORR
Description: The ORR was defined as percentage of participants with a BOR characterized as either a CR or PR, recorded from randomization until documented PD or death relative to the total number of participants. ORR analysis was based on BOR assessed by BICR using RECIST v1.1. Per RECIST v1.1, CR is disappearance of all target lesions; PR is >=30% decrease in the sum of the longest diameter of target lesions; and overall response = CR + PR. Per protocol, participants had CT-scans and brain MRI every 6 weeks to measure tumor lesion size. This was continued throughout treatment until PD or commencement of new anti-neoplastic therapy.
Time Frame: as for outcome 7
Population: Part 2: The ITT population included all randomized participants.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Part 2: Irinotecan Liposome Injection 70 mg/m^2 | Part 2: Topotecan 1.5 mg/m^2
Number analyzed (Participants) | 229 | 232
percentage of participants | 44.1 [37.57 to 50.79] | 21.6 [16.44 to 27.41]
Statistical Analysis 1: Comparison: Part 2: Irinotecan Liposome Injection 70 mg/m^2 vs Part 2: Topotecan 1.5 mg/m^2; Test type: Other; p < 0.0001, Cochran-Mantel-Haenszel — ORR difference, 95% CI and P-value are obtained from the Cochran-Mantel-Haenszel test stratified by corrected region and corrected platinum sensitivity; Difference in ORR = 22.29, 95% CI 2-sided [13.97 to 30.61]

9. Secondary Outcome: Part 2: Median Duration of Response (DoR)
Description: The DoR was defined as time from the first documented objective response (CR or PR, whichever was earlier) to the date of first documented PD or death due to any cause. The DoR analysis was based on BOR assessed by BICR using RECIST v1.1. Per RECIST v1.1, CR is disappearance of all target lesions and PR is >=30% decrease in the sum of the longest diameter of target lesions. The DoR was calculated using Kaplan-Meier technique. Per protocol, participants had CT-scans and brain MRI every 6 weeks to measure tumor lesion size. This was continued throughout treatment until PD or commencement of new anti-neoplastic therapy.
Time Frame: as for outcome 7
Population: Part 2: The ITT population included all randomized participants. Only participants with objective response were analyzed.
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Part 2: Topotecan 1.5 mg/m2 IV: Eligible participants received topotecan 1.5 mg/m2 i.v. over 30 minutes daily for 5 consecutive days, starting on Day 1 of a 21-day cycle for 6 weeks.
Arm/Group | Part 2: Irinotecan Liposome Injection 70 mg/m^2 | Part 2: Topotecan 1.5 mg/m2 IV
Number analyzed (Participants) | 101 | 50
months | 4.14 [3.06 to 4.34] | 4.17 [2.86 to 4.76]

10. Secondary Outcome: Part 2: Median Time to Objective Response (OR)
Description: Time to OR as per RECIST v1.1 criteria according to BICR was defined as time from the date of randomization to the date of first documented objective tumor response (CR or PR, whichever was first). Per RECIST v1.1, CR is disappearance of all target lesions; PR is >=30% decrease in the sum of the longest diameter of target lesion. Participants with a new anti-cancer therapy prior to OR were censored at the last tumor assessment prior to new anti-cancer therapy. Per protocol, participants had CT-scans and brain MRI every 6 weeks to measure tumor lesion size. This was continued throughout treatment until PD or commencement of new anti-neoplastic therapy.
Time Frame: as for outcome 7
Population: as for outcome 9
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Part 2: Irinotecan Liposome Injection 70 mg/m^2 | Part 2: Topotecan 1.5 mg/m^2
Number analyzed (Participants) | 101 | 50
months | 1.68 [1.51 to 4.11] | 12.65 [8.41 to NA] — Upper limit of CI was not estimable due to insufficient number of participants with events at study closure.

11. Secondary Outcome: Change From Baseline in European Organization for Research and Treatment of Cancer Quality of Life Questionnaire - Core 30 (EORTC QLQ-C30)/Lung Cancer Supplement (LC13) Dyspnea Scale at Week 12
Description: The EORTC QLQ-LC13 is a lung cancer specific module used in conjunction with EORTC QLQ-C30 and covers typical symptoms of lung cancer (cough, pain, dyspnea, sore mouth, peripheral neuropathy, hair loss). Scores range from 0-100 and a high score represents a high level of symptomatology/problems/worse QoL. Baseline was defined as the last non-missing measurement taken prior to reference start date. Change from baseline in dyspnea scale was calculated regardless of premature study treatment discontinuation. Participants completed these questionnaires on an electronic tablet every 6 weeks during treatment and it was continued until PD or commencement of new anti-neoplastic therapy.
Time Frame: Baseline (Day 1) and Week 12
Population: Part 2: The ITT population included all randomized participants. Only participants analyzed at Week 12 are reported.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Part 2: Irinotecan Liposome Injection 70 mg/m^2 | Part 2: Topotecan 1.5 mg/m^2
Number analyzed (Participants) | 106 | 114
scores on a scale | 4.6 (20.74) | 1.9 (19.17)

12. Secondary Outcome: Change From Baseline in EORTC QLQ-LC13 Cough Scale at Week 12
Description: The EORTC QLQ-LC13 is a lung cancer specific module used in conjunction with EORTC QLQ-C30 and covers typical symptoms of lung cancer (cough, pain, dyspnea, sore mouth, peripheral neuropathy, hair loss). Score ranges from 0-100 scale and a high score represents a high level of symptomatology/problems/worse QoL. Baseline was defined as the last non-missing measurement taken prior to reference start date. Change from baseline in cough scale was calculated regardless of premature study treatment discontinuation. Participants completed these questionnaires on an electronic tablet every 6 weeks during treatment and it was continued until PD or commencement of new anti-neoplastic therapy.
Time Frame: Baseline (Day 1) and Week 12
Population: Part 2: The ITT population included all randomized participants. Only participants analyzed at Week 12 are reported.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Part 2: Irinotecan Liposome Injection 70 mg/m^2 | Part 2: Topotecan 1.5 mg/m^2
Number analyzed (Participants) | 106 | 114
scores on a scale | 1.6 (25.77) | -1.2 (27.31)

ADVERSE EVENTS:
Time Frame: The TEAEs were reported from the time of first study treatment administration (Day 1) up to 30 days after the date of last study treatment administration, approximately 680 days for Part 1 and 1452 days for Part 2. All-Cause Mortality: approximately 1919 days
Description: Part 1: Safety population included all enrolled participants who were treated with at least 1 dose of irinotecan liposome injection. Part 2: Safety population included all randomized participants who were treated with at least 1 dose of study treatment. AEs are coded using MedDRA version 26.0. During all study visits, participants were asked to report any adverse events/symptoms since prior study visit.
Arm/Group | Part 1: Irinotecan Liposome Injection 85 mg/m^2 | Part 1: Irinotecan Liposome Injection 70 mg/m^2 | Part 2: Irinotecan Liposome Injection 70 mg/m^2 | Part 2: Topotecan 1.5 mg/m^2
All-Cause Mortality (participants affected / at risk) | 5/5 | 23/25 | 201/226 | 205/223
Serious Adverse Events (participants affected / at risk) | 4/5 | 9/25 | 106/226 | 88/223
Other Adverse Events (participants affected / at risk) | 5/5 | 25/25 | 212/226 | 220/223
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 1: Irinotecan Liposome Injection 85 mg/m^2 (N=5) | Part 1: Irinotecan Liposome Injection 70 mg/m^2 (N=25) | Part 2: Irinotecan Liposome Injection 70 mg/m^2 (N=226) | Part 2: Topotecan 1.5 mg/m^2 (N=223)
Cardiac arrest (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cardiac tamponade (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Coronary artery disease (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pericardial effusion (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ectopic antidiuretic hormone secretion (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (2) | 1 (1) | 19 (25) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 2 (2) | 3 (3)
Oesophageal stenosis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (2) | 0 (0) | 3 (3) | 3 (3)
Enterocolitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 4 (4) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Duodenal ulcer perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Enteritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ileus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Narcotic bowel syndrome (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pancreatitis acute (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hepatotoxicity (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Liver disorder (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hepatitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Biliary obstruction (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 2 (2) | 2 (2) | 16 (18) | 7 (8)
Abdominal sepsis (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 13 (16) | 8 (9)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 5 (6) | 2 (2)
Suspected COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 6 (7) | 2 (2)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
COVID-19 pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Atypical pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Clostridium difficile infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Erysipelas (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Infectious pleural effusion (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonia viral (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Liver function test abnormal (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 8 (16)
Neutrophil count decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood creatinine increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Transaminases increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
White blood cell count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (3)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1) | 5 (11)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Embolism arterial (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Superior vena cava syndrome (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Embolism (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haemorrhage (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Subclavian vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 2 (2) | 19 (24)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 5 (5) | 13 (13)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 13 (21)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 2 (2) | 9 (10)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 6 (7)
Myelosuppression (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Asthenia (General disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Death (General disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Multiple organ dysfunction syndrome (General disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Complication associated with device (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
General physical health deterioration (General disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Anaphylactic reaction (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypersensitivity (Immune system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Overdose (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 5 (6) | 0 (0)
Radiation pneumonitis (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Exposure to SARS-CoV-2 (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Procedural pneumothorax (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Myopathy (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cerebral infarction (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (2)
Haemorrhage intracranial (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Seizure (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Cerebral ischaemia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Myoclonus (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vertebrobasilar stroke (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Confusional state (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Cystitis haemorrhagic (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Renal failure (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Renal impairment (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 7 (7) | 3 (3)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (2) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Aortic thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Device related thrombosis (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 1: Irinotecan Liposome Injection 85 mg/m^2 (N=5) | Part 1: Irinotecan Liposome Injection 70 mg/m^2 (N=25) | Part 2: Irinotecan Liposome Injection 70 mg/m^2 (N=226) | Part 2: Topotecan 1.5 mg/m^2 (N=223)
Anaemia (Blood and lymphatic system disorders) | 2 (7) | 7 (11) | 82 (193) | 177 (773)
Neutropenia (Blood and lymphatic system disorders) | 3 (3) | 4 (7) | 41 (124) | 137 (532)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 4 (11) | 11 (20) | 131 (487)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 29 (82) | 94 (397)
Lymphopenia (Blood and lymphatic system disorders) | 1 (3) | 1 (5) | 22 (54) | 27 (133)
Coagulopathy (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 2 (4) | 2 (2) | 3 (3)
Adrenal insufficiency (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Visual impairment (Eye disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 5 (17) | 22 (80) | 128 (393) | 43 (70)
Nausea (Gastrointestinal disorders) | 3 (5) | 11 (17) | 96 (170) | 58 (94)
Vomiting (Gastrointestinal disorders) | 1 (5) | 9 (16) | 47 (83) | 27 (46)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 5 (5) | 41 (56) | 8 (8)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 5 (5) | 11 (12) | 8 (10)
Constipation (Gastrointestinal disorders) | 2 (3) | 3 (4) | 29 (42) | 35 (46)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 3 (3) | 5 (6) | 5 (6)
Stomatitis (Gastrointestinal disorders) | 1 (1) | 2 (4) | 6 (7) | 6 (12)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 0 (0) | 7 (8) | 2 (2)
Flatulence (Gastrointestinal disorders) | 1 (1) | 0 (0) | 4 (4) | 0 (0)
Asthenia (General disorders) | 1 (4) | 10 (22) | 60 (111) | 50 (90)
Fatigue (General disorders) | 1 (3) | 4 (10) | 48 (83) | 43 (58)
Non-cardiac chest pain (General disorders) | 0 (0) | 3 (3) | 14 (19) | 18 (19)
Oedema peripheral (General disorders) | 1 (1) | 2 (4) | 12 (15) | 7 (8)
Pyrexia (General disorders) | 0 (0) | 3 (4) | 10 (11) | 16 (18)
Pain (General disorders) | 1 (1) | 0 (0) | 6 (7) | 4 (4)
Urinary tract infection (Infections and infestations) | 0 (0) | 3 (4) | 6 (6) | 3 (3)
Herpes zoster (Infections and infestations) | 1 (1) | 1 (1) | 2 (2) | 4 (5)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 2 (2) | 1 (2) | 5 (5)
Weight decreased (Investigations) | 1 (2) | 9 (11) | 65 (112) | 26 (43)
Alanine aminotransferase increased (Investigations) | 1 (3) | 5 (8) | 35 (59) | 22 (30)
Gamma-glutamyltransferase increased (Investigations) | 1 (2) | 4 (7) | 10 (17) | 6 (6)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 3 (5) | 27 (41) | 14 (17)
Blood alkaline phosphatase increased (Investigations) | 1 (2) | 3 (4) | 19 (29) | 14 (18)
Platelet count decreased (Investigations) | 0 (0) | 0 (0) | 9 (34) | 59 (220)
Neutrophil count decreased (Investigations) | 0 (0) | 0 (0) | 21 (46) | 45 (115)
White blood cell count decreased (Investigations) | 0 (0) | 0 (0) | 22 (46) | 34 (102)
Blood creatinine increased (Investigations) | 0 (0) | 0 (0) | 19 (30) | 9 (21)
Blood lactate dehydrogenase increased (Investigations) | 0 (0) | 1 (1) | 11 (16) | 13 (23)
Decreased appetite (Metabolism and nutrition disorders) | 4 (5) | 10 (17) | 81 (120) | 43 (56)
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 (2) | 9 (13) | 19 (46) | 19 (30)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 7 (10) | 36 (53) | 15 (29)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 3 (5) | 13 (15) | 4 (4)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 3 (3) | 17 (21) | 15 (23)
Hypocalcaemia (Metabolism and nutrition disorders) | 1 (1) | 2 (2) | 17 (26) | 5 (12)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 2 (2) | 24 (43) | 24 (61)
Hyperuricaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 13 (18) | 11 (14)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 23 (40) | 13 (25)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 8 (8) | 13 (15) | 12 (13)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1) | 11 (13) | 16 (19)
Dizziness (Nervous system disorders) | 0 (0) | 4 (4) | 12 (14) | 20 (24)
Headache (Nervous system disorders) | 1 (1) | 2 (2) | 11 (13) | 13 (16)
Somnolence (Nervous system disorders) | 0 (0) | 2 (2) | 3 (3) | 2 (2)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1) | 11 (14) | 15 (15)
Renal failure (Renal and urinary disorders) | 1 (1) | 3 (3) | 2 (2) | 2 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 4 (7) | 19 (24) | 27 (35)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (4) | 15 (18) | 19 (23)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (2)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 16 (20) | 27 (34)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 3 (9) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 5 (8) | 6 (8)
Hypotension (Vascular disorders) | 1 (1) | 3 (3) | 10 (10) | 7 (10)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 2 (2) | 2 (2) | 3 (3)
Diverticulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2021-10-07): https://cdn.clinicaltrials.gov/large-docs/13/NCT03088813/Prot_000.pdf
  • Statistical Analysis Plan (2021-11-11): https://cdn.clinicaltrials.gov/large-docs/13/NCT03088813/SAP_001.pdf